CLINICAL TRIAL: NCT00464776
Title: A Randomized, Double-blind, Cross-over, 4-period, 4 Treatment, Within-subject Placebo-controlled Study to Assess the Optimal Renoprotective Dose of Aliskiren in Hypertensive Type 2 Diabetic Patients With Incipient or Overt Nephropathy
Brief Title: Study to Assess the Optimal Renoprotective Dose of Aliskiren in Hypertensive Patients With Type 2 Diabetes and Incipient or Overt Nephropathy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSPP100A2240
Record Dates: First submitted 2007-04-21; First posted 2007-04-24 (Estimated); Last update posted 2011-02-04 (Estimated); Status verified 2011-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Randomized; double-blind; cross-over; 4-period; 4 treatment; within-subject placebo-controlled study; assess optimal renoprotective dose of Aliskiren; hypertensive type 2 diabetes patients; incipient or overt nephropathy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — aliskiren

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): Various sequences of 3 doses of Aliskiren plus placebo
  Interventions: Drug: Aliskiren
- 2 (Experimental): Various sequences of 3 doses of Aliskiren plus placebo
  Interventions: Drug: Aliskiren
- 3 (Experimental): Various sequences of 3 doses of Aliskiren plus placebo
  Interventions: Drug: Aliskiren
- 4 (Experimental): Various sequences of 3 doses of Aliskiren plus placebo
  Interventions: Drug: Aliskiren

INTERVENTIONS:
Drug: Aliskiren
  Other Names: SPP100
  Arms: 1
Drug: Aliskiren
  Other Names: SPP100
  Arms: 2
Drug: Aliskiren
  Other Names: SPP100
  Arms: 3
Drug: Aliskiren
  Other Names: SPP100
  Arms: 4

SUMMARY:
This study will assess the optimal renoprotective dose of Aliskiren in hypertensive type 2 diabetes patients with incipient or overt nephropathy

ELIGIBILITY:
Inclusion Criteria:

* Male and/or female patients from 30-80 years of age.
* Type 2 diabetes (defined using World Health Organization criteria)
* Incipient or overt nephropathy (urinary albumin excretion 100 but ≤ 2000 mg/day).
* Glomerular filtration rate (GFR) 40ml per minute
* To be eligible for randomization, patients must fulfill the following criteria:

  1. Patients on ongoing hypertensive therapy must have a blood pressure ≥ 135/85 mm Hg but lower than 170/105 mm Hg at Visit 3 (Day -1, Period 1) AND patients must be on stable antihypertensive medications for at least 8 weeks prior to Visit 2 (Run-in period)
  2. Newly diagnosed hypertensive patients must have a blood pressure ≥ 135/85 mm Hg but lower than 170/105 mm Hg at Visit 3 (Day -1, Period 1)
* Female patients must be postmenopausal or must have had a bilateral oophorectomy or must have been surgically sterilized or hysterectomized at least 6 months prior to screening
* Oral body temperature within the range 35.0-37.5 °C
* Able to provide written informed consent prior to study participation.
* Able to communicate well with the investigator and comply with the requirements of the study.
* Patients must be willing and medically able to discontinue anti-hypertensive treatment or any other medication which is prohibited in the study protocol.
* Patients must be on stable hypoglycemic medications for at least 8 weeks prior to visit 1 (Screening visit).

Exclusion Criteria:

* Use of any prescription drug or over-the-counter (OTC) medication which is prohibited by the protocol.
* Severe Hypertension Grade 3 WHO classification Mean Sitting Diastolic Blood Pressure (MSDBP) 110 mmHg and/or Mean Sitting Systolic Blood Pressure MSSBP 180 mmHg)
* Acetylsalicyclic acid (ASA) treatment >1g/day or regular use of Non steroidal anti-inflammatory drugs (NSAIDs)
* Kidney disease not caused by diabetes or hypertension
* Serum potassium < 3.5 or > 5.1 mEq/L
* GFR < 40 ml/min/1.73m2 as measured by the Modification of Diet in Renal Disease (MDRD) formula
* Serum albumin < 2.0mg/dL
* History of hypertensive encephalopathy or cerebrovascular accident at any time prior to Visit 1
* Transient ischemic cerebral attack during the 6 months prior to Visit 1
* Current diagnosis of heart failure New York Heart Association (NYHA) Class II-IV
* History of myocardial infarction, unstable angina pectoris, coronary bypass surgery, or any percutaneous coronary intervention (PCI) during the 6 months prior to Visit 1
* Second or third degree heart block without a pacemaker
* Concurrent potentially life threatening arrhythmia or symptomatic arrhythmia
* Clinically significant valvular heart disease
* Type 1 diabetes mellitus
* Uncontrolled Type II diabetes mellitus Hemoglobin subtype A1C (HbA1C) >11 %
* History of malignancy including leukemia and lymphoma (but not basal cell skin carcinoma) within the past five years
* Pregnant or nursing women
* Participation in any clinical investigation within 4 weeks prior to dosing or longer if required by local regulation.
* Donation or loss of 400 mL or more of blood within 8 weeks prior to dosing.
* Significant illness within the two weeks prior to dosing.
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of study drugs including, but not limited to, any of the following:

  * History of major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, or bowel resection
  * Currently active or previously active inflammatory bowel disease during the 12 months prior to Visit 1
  * Currently active gastritis, duodenal or gastric ulcers, or gastrointestinal/rectal bleeding during the 3 months prior to Visit 1.
  * Any history of pancreatic injury, pancreatitis or evidence of impaired pancreatic function/injury as indicated by abnormal lipase or amylase
  * Evidence of hepatic disease, a history of hepatic encephalopathy, a history of esophageal varices, or a history of portocaval shunt
  * Current treatment with cholestyramine or cholestipol resins
* History of immunocompromise, including a positive HIV test result.
* History of a positive Hepatitis B surface antigen (HBsAg) or Hepatitis C test result.
* History of drug or alcohol abuse within the 12 months prior to dosing.
* Persons directly involved in the execution of this protocol.
* Any condition that in the opinion of the investigator or the Novartis medical monitor would jeopardize the evaluation of efficacy or safety
* History of noncompliance to medical regimens or unwillingness to comply with the study protocol
* Known or suspected contraindications to the study medications, including history of allergy to ACE inhibitors and/or to thiazide diuretics or other sulfonamide derived drug
* Any surgical or medical condition, which in the opinion of the investigator, may place the patient at higher risk from his/her participation in the study, or is likely to prevent the patient from complying with the requirements of the study or completing the study
* Patients who previously participated in any Aliskiren study.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2005-10; Primary Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Investigate the antiproteinuric effect of increasing doses of Aliskiren compared to matching placebo. | End of study

SECONDARY OUTCOMES:
Assess the effect on Glomerular Filtration Rate (GFR) of multiple dose administration of Aliskiren. | End of study
Assess the effect on blood pressure of multiple dose administration of Aliskiren. | End of study
To investigate whether there is a change in biomarkers of inflammation and cardiovascular risk. | End of study

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Investigative site
Locations (1):
- Novartis, Gentofte Municipality, Denmark

REFERENCES:
- [Derived] Persson F, Rossing P, Reinhard H, Juhl T, Stehouwer CD, Schalkwijk C, Danser AH, Boomsma F, Frandsen E, Parving HH. Optimal antiproteinuric dose of aliskiren in type 2 diabetes mellitus: a randomised crossover trial. Diabetologia. 2010 Aug;53(8):1576-80. doi: 10.1007/s00125-010-1789-6. Epub 2010 May 18. PMID 20480132